CLINICAL TRIAL: NCT02690987
Title: Do Appetitive Gut Hormones Reduce Addictive and Eating Behaviours in Obesity, and Nicotine and Alcohol Dependence?
Brief Title: Gut Hormones in Obesity, Nicotine and Alcohol Dependence
Acronym: GHADD
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 15/LO/1041; MR/M007022/1 (Other Grant/Funding Number: UK Medical Research Council)
Record Dates: First submitted 2015-11-11; First posted 2016-02-24 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Obesity; Smoking Cessation; Alcoholism
Keywords: tobacco; GLP1; ghrelin; alcohol; appetite; reward; addiction; hormone; cigarette; functional MRI
MeSH Terms: conditions — Obesity; Smoking Cessation; Alcoholism; Behavior, Addictive | interventions — Exenatide; ghrelin, des-n-octanoyl; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Overweight/obese subjects (Experimental): Overweight/obese volunteers with BMI 28.0-50.0 kg/m2, otherwise healthy. This group will receive interventions with saline as placebo, Exenatide and desacyl ghrelin infusions at separate visits in a within subject randomised crossover design.
  Interventions: Drug: Exenatide; Biological: Desacyl ghrelin; Biological: Saline
- Ex-smokers (Experimental): Abstinent tobacco dependent individuals who score at least moderately on tobacco dependence as measured retrospectively using the Fagerström Test for Nicotine Dependence (FTND), and who have been in stable tobacco abstinence for at least 6 weeks.
  This group will receive interventions with saline as placebo, Exenatide and desacyl ghrelin infusions at separate visits in a within subject randomised crossover design.
  Interventions: Drug: Exenatide; Biological: Desacyl ghrelin; Biological: Saline
- Ex-alcohol dependent subjects (Experimental): Abstinent alcohol dependent individuals who score at least moderately alcohol dependent as measured retrospectively using the Severity of Alcohol Dependence Questionnaire (SADQ), and who have been abstinent for at least 6 weeks.
  This group will receive interventions with saline as placebo, Exenatide and desacyl ghrelin infusions at separate visits in a within subject randomised crossover design.
  Interventions: Drug: Exenatide; Biological: Desacyl ghrelin; Biological: Saline

INTERVENTIONS:
Drug: Exenatide — Exenatide is a commercially available GLP-1 receptor agonist. It is a synthetic form of exendin-4, a protein extracted from the saliva of a Gila monster lizard, which exhibits 53% sequence identity to human GLP-1.
  The planned intravenous Exenatide infusion dose is expected to be 0.06 pmol/kg/min aiming for maintenance plasma concentrations of ~130-190 pg/mL.
  Other Names: Byetta
Biological: Desacyl ghrelin — Ghrelin is a 28 amino acid stomach-derived peptide hormone, with the desacyl ghrelin (DAG) form inactive at the GHSR1a receptor. Good Manufacturing Practice (GMP)-grade DAG is obtained from Clinalfa (Bachem AG, Bubendorf, Switzerland).
  The planned intravenous DAG infusion dose is expected to be 4.0 mcg/kg/hour aiming for maintenance plasma concentrations of ~13-19 ng/mL.
  Other Names: Unacylated ghrelin
Biological: Saline — The placebo visit will involve an intravenous infusion of normal saline.

SUMMARY:
The "Gut Hormones in Addiction" study is a proof-of-concept experimental medicine human study to answer the following questions:

1. Does the administration of the hormone desacyl ghrelin reduce core behavioural components of addiction in dependent individuals who have recently stopped smoking tobacco or drinking alcohol, or overweight/obese subjects?
2. Does the administration of the drug Exenatide reduce core behavioural components of addiction in dependent individuals who have recently stopped smoking tobacco or drinking alcohol, or overweight/obese subjects?
3. Does the administration of desacyl ghrelin or Exenatide reduce reward responses to high-calorie foods and appetite in dependent individuals who have recently stopped smoking tobacco or drinking alcohol, or overweight/obese subjects?

DETAILED DESCRIPTION:
Obesity, smoking and alcohol dependence are major health burdens to society. Relapse after alcohol and smoking abstinence is common despite the use of combined behavioural support and current limited available medications. In obesity, nonsurgical interventions have also been disappointing in achieving longterm weight loss. Therefore, there is a pressing need to develop novel drug treatments for addiction derived from knowledge of brain mechanisms related to relapse and reward responses to food and drugs.

There is evidence in animals that some gut hormones, produced in the stomach and intestine, influence the consumption of food and desire for food, but also alcohol, nicotine and other drugs of abuse. Examples of such gut hormones are glucagon-like peptide1 (GLP1) and ghrelin.

The influence of these hormones is exerted through brain systems involved in the core behavioural components of addiction: reward sensitivity, stress, impulsivity and compulsivity. These components are often also seen in obesity and food-related disorders such as binge eating disorder. It is unknown whether these gut hormones directly influence the core behavioural components of addiction in humans, particularly during abstinence.

The investigators will examine the acute effects of Exenatide (mimics GLP1) and desacyl ghrelin (counteracts active acyl ghrelin), which are infused through a vein, on brain reward systems, craving for food, cigarettes and alcohol, and addictive and eating behaviours.

The investigators will recruit adults with nicotine or alcohol dependence who have recently stopped smoking or drinking, and overweight/obese adults. The investigators will use functional magnetic resonance imaging (MRI) brain scans and computer-based test over 3 separate study days to study different aspects of eating and addictive behaviours.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female volunteers between the ages of 18 and 60 years.
2. Healthy as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests, cardiac monitoring and a psychiatric evaluation. Any volunteer with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included, only if the investigators concur that the finding is unlikely to jeopardize either volunteer safety or study integrity.
3. The subject is capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
4. The subject is able to read, comprehend and record information written in English.
5. For non-dependent groups:

   i) Overweight/obese volunteers with BMI 28.0-50.0 kg/m2.
6. For addiction groups:

Subjects meeting Diagnostic and Statistical Manual (DSM)-V criteria for previous nicotine or alcohol dependence, but who are in early stable abstinence (>6 weeks). Minor lapses within this time period will be allowed but not relapses into dependence.

ii) Abstinent alcohol dependent individuals who score at least moderately alcohol dependent as measured retrospectively using the Severity of Alcohol Dependence Questionnaire (SADQ), and who have been abstinent for >6 weeks.

iii) Abstinent tobacco dependent individuals who score at least moderately on tobacco dependence as measured retrospectively using the Fagerström Test for Nicotine Dependence (FTND), and who have been in stable tobacco abstinence for >6 weeks.

Exclusion Criteria:

Potential volunteers will NOT be eligible for inclusion in this study if any of the following criteria apply:

1. Previous history of recreational use or abuse of other substances of addiction will be permissible, but there should be no use of any illegal drugs (except cannabis) in the month prior to the Screening Visit or during the course of the study, except where specified for individual groups below.
2. For individual groups:

   i) Overweight/obese group: history of or current alcohol abuse or dependence; nicotine use other than "never smoked", i.e. >100 cigarettes lifetime use; history of dependence, abuse or heavy recreational use of cocaine, cannabis, opiates or other substance of abuse; history of problem gambling. Any previous or current psychiatric diagnosis listed in Diagnostic and Statistical Manual (DSM)-V Axis I, which in the opinion of the clinical team will compromise conduct and interpretability of the study.

   ii) Abstinent tobacco dependent group: history of or current alcohol abuse or dependence; current dependence for cocaine, cannabis, opiates or other substance of abuse, or problem gambling (previous history will be allowed); taking varenicline, bupropion or other prescription medications for smoking cessation. Any previous or current psychiatric diagnosis listed in Diagnostic and Statistical Manual (DSM)-V Axis I, which in the opinion of the clinical team will compromise conduct and interpretability of the study.

   iii) Abstinent alcohol dependent group: current dependence for cocaine, cannabis, opiates or other substance of abuse, or problem gambling (previous history will be allowed); taking prescription medication for alcohol or smoking cessation or withdrawal; smoking is allowed past or present including dependence; current nicotine replacement therapy is allowed.
3. Currently suffering from Diagnostic and Statistical Manual (DSM)-V depressive disorder or on anti-depressant medication, though a history of depression or anxiety will be allowed. A current or past history of enduring severe mental illness (e.g., schizophrenia, bipolar affective disorder) will not be allowed.

   For all groups:
4. Cannabis use up to five times in the month prior to the Screening Visit will be allowed, but no use within one week of experimental assessments; no use of any other illegal drugs in the month prior to the Screening Visit or during the course of the study.
5. Intoxication at any of the visits, as manifested by difficulty in walking, slurring of speech, difficulty concentrating or drowsiness (or by the subject volunteering this information directly to the research team).
6. Positive drug/alcohol screens on testing at the screening visit, other than that explicable by other causes (e.g. recent use of opiate containing analgesic etc), at the discretion of the research team.
7. Carbon monoxide levels of =/>10ppm in the overweight/obese and abstinent smoker groups at screening visit.
8. Use of current regular prescriptions (including smoking or alcohol cessation medicines such as Disulfiram, Acamprosate, Naltrexone, Bupropion; weight loss medication including Orlistat, Metformin, GLP-1 agonists, Bupropion, Naltrexone), or over-the-counter medications that in the opinion of the Investigators may affect subject safety or outcome measures.
9. Pulse rate <40 or >100 beats per minute OR systolic blood pressure >160 and <100 and a diastolic blood pressure >95 and <50 in the semi-supine position.
10. Claustrophobia or feels that they will be unable to lay still on their back in the MRI scanner for a period of ~80 minutes.
11. Presence of a cardiac pacemaker or other electronic device or ferromagnetic metal foreign bodies as assessed by a standard pre-MRI questionnaire and radiographer.
12. History or presence of a neurological diagnosis (not limited to but including, for example, stroke, epilepsy, space occupying lesions, multiple sclerosis, Parkinson's disease, vascular dementia, transient ischemic attack, that may influence the outcome or analysis of the scan results). A history of alcohol-related or alcohol-withdrawal seizures will be allowed for volunteers in the abstinent alcoholic group.
13. Significant current or past medical or psychiatric history that, in the opinion of the investigators, contraindicates their participation.
14. Clinically significant head injury (e.g. requiring hospitalisation or surgical intervention) that in the opinion of the investigators may affect subject safety or outcome measures.
15. Unwillingness or inability to follow the procedures outlined in the protocol.
16. Any of the following liver function tests (LFT) abnormalities at screening: Alkaline Phosphatase, aspartate aminotransferase (AST), alanine aminotransferase (ALT) or gammaGT > 4 x upper limit of normal (ULN), International Normalised ratio (INR) > 1.5, Albumin <25 g/L, raised bilirubin (other than just isolated i.e. without other liver function tests abnormalities).
17. History of decompensated alcoholic liver disease - i.e. history of variceal bleeding, ascites, jaundice, encephalopathy.
18. History of pancreatitis from any cause.
19. History of type 1 or type 2 diabetes mellitus.
20. ECG abnormality, which in the opinion of the study physician, is clinically significant and represents a safety risk.
21. The volunteer has participated in a clinical trial and has received an investigational product within the following time period prior to the first experimental visit in the current study: 90 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
22. Exposure to more than 3 new investigational medicinal products within 12 months prior to the scan.
23. History of sensitivity to any of the peptides, or components thereof, or a history of drug or other allergy that, in the opinion of the investigators, contraindicates their participation.
24. Diagnosis of endocrine disorder, including uncontrolled hypothyroidism (stable treated hypothyroidism with currently normal thyroid function tests is allowed), history of hyperthyroidism or Cushing's syndrome, which, in the opinion of the investigators, may affect subject safety or outcome measures.
25. History of ischaemic heart disease, heart failure, cardiac arrhythmia or peripheral vascular or cerebrovascular disease.
26. History or presence of significant respiratory, gastrointestinal, hepatic, oncological or renal disease or other condition that in the opinion of the Investigators may affect subject safety or outcome measures.
27. Previous bariatric surgery for obesity including Roux-en-Y gastric bypass, gastric banding, sleeve gastrectomy.
28. Current pregnancy or breast-feeding in female volunteers.
29. Vegetarian, vegan, gluten or lactose-intolerant.
30. Volunteers who have donated, or intend to donate, blood within three months before the screening visit or following study visit completion.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-08-21 (Actual); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Functional MRI measure of brain activation during cigarette, alcohol and food picture evaluation task | 4 years
  Blood oxygen level dependent (BOLD) signal in brain reward systems to cigarette, alcohol and food pictures vs. object pictures

SECONDARY OUTCOMES:
Functional MRI measure of brain activation during anticipation of winning monetary reward (monetary incentive delay task) | 4 years
  Blood oxygen level dependent (BOLD) signal in striatum to anticipation of winning vs. not winning money
Functional MRI measure of brain activation during negative emotional reactivity task | 4 years
  Blood oxygen level dependent (BOLD) signal in amygdala during viewing of evocative vs. neutral pictures
Functional MRI measure of brain activity in salience resting state network | 4 years
  Network integrity of blood oxygen level dependent (BOLD) signal in salience resting state network
Functional MRI measure of brain activity in limbic resting state network | 4 years
  Network integrity of blood oxygen level dependent (BOLD) signal in limbic resting state network
Functional MRI measure of brain activity in default mode resting state network | 4 years
  Network integrity of blood oxygen level dependent (BOLD) signal in default mode resting state network

OTHER OUTCOMES:
Hunger visual analogue scale rating | 4 years
  Appetite measure
Alcohol Urge Questionnaire | 4 years
  Alcohol craving measure
Questionnaire of Smoking Urges | 4 years
  Cigarette craving measure
Food craving visual analogue scale rating | 4 years
Progressive ratio task breakpoint | 4 years
  Measure of motivation to obtain sweet palatable food
Percentage of unsuccessful stop trials | 4 years
  Motor response inhibition measure
Energy intake at test meal in kilocalories | 4 years
Energy intake of sugar at test meal as percentage of total | 4 years
Energy intake of fat at test meal as percentage of total | 4 years
Ratio of speed of approach to avoidance for food vs. object pictures | 4 years
Ratio of speed of approach to avoidance for alcohol vs. object pictures | 4 years
Ratio of speed of approach to avoidance for cigarette vs. object pictures | 4 years
Food picture appeal rating | 4 years
Alcohol picture appeal rating | 4 years
Cigarette picture appeal rating | 4 years
Plasma glucose concentration | 4 years
Serum insulin concentration | 4 years
Serum cortisol concentration | 4 years
Serum growth hormone concentration | 4 years
Plasma GLP1 concentration | 4 years
Plasma peptide YY concentration | 4 years
Plasma exenatide concentration | 4 years
Plasma desacyl ghrelin concentration | 4 years
Plasma acyl ghrelin concentration | 4 years
Nausea visual analogue scale rating | 4 years
Fullness visual analogue scale rating | 4 years
Sweet taste intensity visual analogue scale rating | 4 years
Fat taste intensity visual analogue scale rating | 4 years
Fat taste just right visual analogue scale rating | 4 years
Sweet taste just right visual analogue scale rating | 4 years
Sweet taste liking visual analogue scale rating | 4 years
Fat taste liking visual analogue scale rating | 4 years
Fat taste pleasant visual analogue scale rating | 4 years
Sweet taste pleasant visual analogue scale rating | 4 years
Paired associates learning task number of trials required to locate patterns correctly | 4 years
  Episodic memory measure
Paired associates learning task memory score | 4 years
  Episodic memory measure
Paired associates learning task number of stages completed | 4 years
  Episodic memory measure
Cambridge gambling task risk taking measure | 4 years
  Neuropsychological test
Cambridge gambling task quality of decision taking measure | 4 years
  Neuropsychological test
Smoking relapse rate at 6 months after completion of the study in ex-smokers | 4 years
Smoking relapse rate at 12 months after completion of the study in ex-smokers | 4 years
Alcohol relapse rate at 6 months after completion of the study in ex-drinkers | 4 years
Alcohol relapse rate at 12 months after completion of the study in ex-drinkers | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Tony Goldstone, MD, PhD, Principal Investigator — Imperial College London; David Nutt, MD, PhD, Principal Investigator — Imperial College London
Locations (1):
- Centre for Neuropsychopharmacology, Division of Brain Sciences, Imperial College London, Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dickson SL, Egecioglu E, Landgren S, Skibicka KP, Engel JA, Jerlhag E. The role of the central ghrelin system in reward from food and chemical drugs. Mol Cell Endocrinol. 2011 Jun 20;340(1):80-7. doi: 10.1016/j.mce.2011.02.017. Epub 2011 Feb 24. PMID 21354264
- [Background] Egecioglu E, Engel JA, Jerlhag E. The glucagon-like peptide 1 analogue Exendin-4 attenuates the nicotine-induced locomotor stimulation, accumbal dopamine release, conditioned place preference as well as the expression of locomotor sensitization in mice. PLoS One. 2013 Oct 18;8(10):e77284. doi: 10.1371/journal.pone.0077284. eCollection 2013. PMID 24204788
- [Background] Goldstone AP, Prechtl CG, Scholtz S, Miras AD, Chhina N, Durighel G, Deliran SS, Beckmann C, Ghatei MA, Ashby DR, Waldman AD, Gaylinn BD, Thorner MO, Frost GS, Bloom SR, Bell JD. Ghrelin mimics fasting to enhance human hedonic, orbitofrontal cortex, and hippocampal responses to food. Am J Clin Nutr. 2014 Jun;99(6):1319-30. doi: 10.3945/ajcn.113.075291. Epub 2014 Apr 23. PMID 24760977
- [Background] Heatherton TF, Kozlowski LT, Frecker RC, Fagerstrom KO. The Fagerstrom Test for Nicotine Dependence: a revision of the Fagerstrom Tolerance Questionnaire. Br J Addict. 1991 Sep;86(9):1119-27. doi: 10.1111/j.1360-0443.1991.tb01879.x. PMID 1932883
- [Background] Saunders JB, Aasland OG, Babor TF, de la Fuente JR, Grant M. Development of the Alcohol Use Disorders Identification Test (AUDIT): WHO Collaborative Project on Early Detection of Persons with Harmful Alcohol Consumption--II. Addiction. 1993 Jun;88(6):791-804. doi: 10.1111/j.1360-0443.1993.tb02093.x. PMID 8329970
- [Background] Shirazi RH, Dickson SL, Skibicka KP. Gut peptide GLP-1 and its analogue, Exendin-4, decrease alcohol intake and reward. PLoS One. 2013 Apr 16;8(4):e61965. doi: 10.1371/journal.pone.0061965. Print 2013. PMID 23613987
- [Background] Tong J, Davis HW, Summer S, Benoit SC, Haque A, Bidlingmaier M, Tschop MH, D'Alessio D. Acute administration of unacylated ghrelin has no effect on Basal or stimulated insulin secretion in healthy humans. Diabetes. 2014 Jul;63(7):2309-19. doi: 10.2337/db13-1598. Epub 2014 Feb 18. PMID 24550190
- [Background] van Bloemendaal L, IJzerman RG, Ten Kulve JS, Barkhof F, Konrad RJ, Drent ML, Veltman DJ, Diamant M. GLP-1 receptor activation modulates appetite- and reward-related brain areas in humans. Diabetes. 2014 Dec;63(12):4186-96. doi: 10.2337/db14-0849. Epub 2014 Jul 28. PMID 25071023
- [Background] Scholtz S, Miras AD, Chhina N, Prechtl CG, Sleeth ML, Daud NM, Ismail NA, Durighel G, Ahmed AR, Olbers T, Vincent RP, Alaghband-Zadeh J, Ghatei MA, Waldman AD, Frost GS, Bell JD, le Roux CW, Goldstone AP. Obese patients after gastric bypass surgery have lower brain-hedonic responses to food than after gastric banding. Gut. 2014 Jun;63(6):891-902. doi: 10.1136/gutjnl-2013-305008. Epub 2013 Aug 20. PMID 23964100